CLINICAL TRIAL: NCT01539330
Title: Assessment of Target Site Pharmacokinetics of Voriconazole in Healthy Volunteers During Sequence Therapy
Acronym: VORTarget-site
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Charlotte Kloft, Head of Department of Clinical Pharmacy, Martin-Luther-Universität Halle-Wittenberg
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KP-VOR03; 2008-008524-32 (EudraCT Number)
Record Dates: First submitted 2012-02-09; First posted 2012-02-27 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: voriconazole; microdialysis; sequence therapy; pharmacokinetics; Target Site Pharmacokinetics
MeSH Terms: interventions — Voriconazole; Microdialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Voriconazole — At beginning of study visit 1 (0-12 h): 6 mg/kg, IV (in the vein) over a period of 120 min
  at beginning of study visit 2 (12-24 h): 6 mg/kg, IV (in the vein) over a period of 120 min
  at beginning of study visit 3 (24-36 h): 4 mg/kg, IV (in the vein) over a period of 80 min
  at beginning of study visit 4 (36-48 h): 4 mg/kg, IV (in the vein) over a period of 80 min
  at beginning of study visit 5 (48-60 h), 6 (60-72 h) and 7 (72-84 h): 200 mg po
  Other Names: VFEND® Pfizer
Other: microdialysis — long-term microdialysis over study days 1-4 (visits 1-7)

SUMMARY:
The present study aims at measuring unbound voriconazole concentrations in plasma and at the relevant target site of systemic fungal infections, i.e. the interstitial space fluid of soft tissues, to assess the target site pharmacokinetics. For this purpose the microdialysis technique will be employed which is capable of measuring the unbound, microbiologically active concentration of antifungals in the interstitial space fluid of virtually all tissues. This is the first human study of this drug employing the microdialysis technique determining the target site concentrations over several days (single and multiple dosing).

DETAILED DESCRIPTION:
Voriconazole, a derivative of fluconazole, is one of the newer triazole antifungal agents launched in 2002. It has demonstrated favourable activity against primary opportunistic fungal pathogens (Aspergillus spp., Candida spp. and Cryptococcus spp.), common dermatophytes and the fungi which cause endemic mycoses. Voriconazole was approved for primary treatment of acute invasive aspergillosis, candidiasis and salvage therapy for rare but serious fungal infections.

Antifungals such as voriconazole should display their pharmacodynamic activity in tissue, more precisely in interstitial space fluid (ISF) of tissue, because this is the site where most of the fungal pathogens are considered to reside. Microdialysis is a novel approach for determination of drug concentration in virtually all tissues and has been used in vivo in animal experiments since 1980s and for about 10 years in human studies. The advantages of this technique are that it is easy to handle and reduces the burden on the patient to a minimum because no tissue extraction is necessary. Microdialysis allows a continuous determination of tissue drug concentrations over a defined time interval. In addition this technique enables to determine only the unbound, i.e. pharmacodynamically active fraction of the extracellular drug concentration at the site of action.

Most pharmacokinetic (PK) data of voriconazole have only been obtained after single dose and only in plasma (bound and unbound concentration). Regarding the pharmacodynamic activity it is more appropriate to determine the unbound concentration at the target site. The novel microdialysis technique allows to evaluate the concentration of voriconazole in subcutaneous interstitial fluid of tissue (unbound concentration), the compartment where most of the pathogens are considered to reside. Apart from multiple i.v. administration of voriconazole, sequence therapy has been introduced, i.e. a switch from direct administration into the systemic circu¬lation to an absorption based administration process, introducing further variability on the PK. A further important reason for assessing voriconazole concentrations during sequence therapy is that the i.v. dose is normalised to body weight but the oral dose is given independently of this demographic dimension.

The study aims at determining unbound voriconazole concentrations in plasma and at the relevant target site of systemic fungal infections, i.e. the interstitial space fluid of soft tissues. Additionally, the PK of voriconazole after single and multiple i.v. and p.o. dosing will be characterised and influencing parameters on the PK will be evaluated.

The design will be a prospective, two part, open-labelled, uncontrolled, study. For this exploratory study no blinding procedure will be performed. Due to the nature of the study, there will be no placebo or comparator arm. The pharmacokinetics will be compared between

* 2 dosing schedules: after single and after multiple dosing
* 2 sampled matrices: plasma and microdialysate

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged between 18 and 50 years
* Body mass index between 20 and 28
* Known genotype of CYP2C19 and CYP2C9
* No regular concomitant (topical or systemic) medication within the last 4 weeks prior to the start of the trial
* Written informed consent given by volunteers after being provided with detailed information about the nature, risks, and scope of the clinical study as well as the expected desirable and adverse effects of the drug
* No legal incapacity and/or other circumstances rendering the subject unable to understand the nature, scope and possible consequences of the study

Exclusion Criteria:

* Known allergy or hypersensitivity against study drug or drug class
* Participation in another clinical study within the last 6 weeks prior to study
* Blood donation within the last 4 weeks prior to study
* Application of live or killed virus or bacteria vaccines within 14 days prior to study
* Alcohol or drug abuse
* Abuse of nicotine
* History of severe allergic or anaphylactic reactions to any medication
* History of or ongoing optic dysfunction (all volunteers will undergo mandatory testing at screening)
* Ongoing bacterial, viral, fungal, or atypical mycobacterial infection
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders
* History of or ongoing hepatic cirrhosis regardless of cause or severity
* History of or ongoing hospital admission for cardiac disease, stroke, or pulmonary disease within the last 5 years
* History of or ongoing symptoms for blood coagulation disorders
* Seropositivity for human immunodeficiency virus (HIV), all volunteers will undergo mandatory testing at screening
* Seropositivity for hepatitis B or C virus (HepB antigen, HepC antibody), all volunteers will undergo testing at screening
* Clinically significant thrombocytopenia, bleeding disorders or a platelet count < 50,000 / µL
* WBC count < 3000/L or > 14,000/L, all volunteers will undergo mandatory testing at screening
* Hepatic enzymes (aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), alkaline phosphatase (AP), gamma-glutamyltranspeptidase (Gamma-GTP), lactate dehydrogenase (LDH)) and bilirubin 3 times the upper limit of normal, all volunteers will undergo mandatory testing at screening
* Serum creatinine 2 times the upper limit of normal, all volunteers will undergo mandatory testing at screening
* Abnormalities in ECG that are considered clinically relevant, all volunteers will undergo mandatory testing at screening
* Unreliability and/or lack of cooperation
* Other objections to participate in the study in the opinion of the investigator

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of voriconazole in plasma and interstitial space fluid of subcutaneous tissue by measuring concentrations of voriconazole in plasma and microdialysate during sequence therapy over 4 days | study day 1-4
  Rich plasma and microdialysate sampling will be done on study day 1,3 and 4. Sparse plasma and microdialysate sampling will be done on study day 2.
  For characterisation of the unbound concentration-time profiles in ultrafiltered plasma and in the interstitial space fluid of subcutaneous adipose tissue (ISF) the following pharmacokinetic (PK) parameters of voriconazole will be determined by suitable PK approaches: Cmax, tmax, AUC, t1/2, CL, V after single dosing and multiple dosing (sequence therapy).

SECONDARY OUTCOMES:
AUC/MIC values | up to 1 year after study visits
  To relate the unbound concentrations in ultrafiltered plasma and interstitial space fluid to reported MIC values in the literature.
genotype analysis | up to 10 weeks before or after study visits
  To exploratory evaluate the genotype of the metabolising enzymes CYP2C9, and CYP2C19 that may have an influence on the pharmacokinetics of voriconazole
cytokine analysis | up to 1 year after study visits
  To exploratory evaluate cytokines as local inflammatory parameters that may have an influence on the pharmacokinetics of voriconazole

CONTACTS AND LOCATIONS:
Overall Officials: Markus Müller, Prof. Dr., Principal Investigator — Medical University of Vienna, Department of Clinical Pharmacology
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Background] Simmel F, Kloft C. Microdialysis feasibility investigations with the non-hydrophilic antifungal voriconazole for potential applications in nonclinical and clinical settings. Int J Clin Pharmacol Ther. 2010 Nov;48(11):695-704. doi: 10.5414/cpp48695. PMID 20979927
- [Result] Simmel F, Kirbs C, Erdogan Z, Lackner E, Zeitlinger M, Kloft C. Pilot investigation on long-term subcutaneous microdialysis: proof of principle in humans. AAPS J. 2013 Jan;15(1):95-103. doi: 10.1208/s12248-012-9412-z. Epub 2012 Oct 13. PMID 23065438